CLINICAL TRIAL: NCT00079352
Title: A Phase I Study of Flavopiridol in Combination With Gemcitabine and Irinotecan in Patients With Metastatic Cancer
Brief Title: Flavopiridol, Gemcitabine, and Irinotecan in Treating Patients With Unresectable or Metastatic Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02580; UNM-0903C; CDR0000355358 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2004-03-08; First posted 2004-03-10 (Estimated); Last update posted 2013-01-25 (Estimated); Status verified 2013-01

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
MeSH Terms: interventions — alvocidib; Gemcitabine; Irinotecan

ARMS (1):
- Treatment (gemcitabine, irinotecan, alvocidib) (Experimental): Patients receive gemcitabine IV over 30 minutes followed by irinotecan IV over 30 minutes on days 1 and 15. Patients also receive flavopiridol IV over 60 minutes on days 2 and 16. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: alvocidib; Drug: gemcitabine hydrochloride; Drug: irinotecan hydrochloride

INTERVENTIONS:
Drug: alvocidib — Given IV
  Other Names: FLAVO; flavopiridol; HMR 1275; L-868275
Drug: gemcitabine hydrochloride — Given IV
  Other Names: dFdC; difluorodeoxycytidine hydrochloride; gemcitabine; Gemzar
Drug: irinotecan hydrochloride — Given IV
  Other Names: Campto; Camptosar; CPT-11; irinotecan; U-101440E

SUMMARY:
This phase I trial is studying the side effects and best dose of flavopiridol when given together with gemcitabine and irinotecan in treating patients with unresectable or metastatic solid tumors. Drugs used in chemotherapy, such as flavopiridol, gemcitabine, and irinotecan, work in different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the maximum tolerated dose and recommended phase II dose of flavopiridol in combination with gemcitabine and irinotecan in patients with unresectable or metastatic solid tumors.

II. Determine the toxicity profile of this regimen in these patients.

OUTLINE: This is a dose-escalation study of flavopiridol.

Patients receive gemcitabine IV over 30 minutes followed by irinotecan IV over 30 minutes on days 1 and 15. Patients also receive flavopiridol IV over 60 minutes on days 2 and 16. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity. Cohorts of 3-6 patients receive escalating doses of flavopiridol until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed solid tumor that is metastatic or unresectable
* Standard curative or palliative measures do not exist or are no longer effective
* No known brain metastases
* Performance status - ECOG 0-2
* Performance status - Karnofsky 60-100%
* More than 12 weeks
* WBC ≥ 3,000/mm^3
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Bilirubin normal
* AST and ALT ≤ 2.5 times upper limit of normal
* Creatinine normal
* Creatinine clearance ≥ 60 mL/min
* No venous thrombosis within the past 6 months
* No thrombotic cerebrovascular accident within the past 6 months
* No myocardial infarction within the past 6 months
* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia
* No ongoing or active infection
* No prior allergic reaction attributed to compounds of similar chemical or biological composition to study agents
* No other concurrent uncontrolled medical condition that would preclude study participation
* No psychiatric illness or social situation that would preclude study participation
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Prior biologic therapy allowed
* More than 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin) and recovered
* Prior endocrine therapy allowed
* More than 4 weeks since prior radiotherapy and recovered
* Prior surgery allowed
* No other concurrent investigational agents
* No concurrent combination antiretroviral therapy for HIV-positive patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2004-04; Primary Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Recommended phase II dose of flavopiridol defined as the highest dose for which no more than one patient develop a >= grade 3 toxicity | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Ian Rabinowitz, Principal Investigator — University of New Mexico
Locations (1):
- University of New Mexico, Albuquerque, New Mexico, United States